CLINICAL TRIAL: NCT01589549
Title: A Phase 2 Trial of Standard of Care Treatment Versus Mesenchymal Stromal Cell Therapy Together With Standard of Care for the Treatment of de Novo Acute Graft Versus Host Disease Following Allogeneic Bone Marrow Transplantation
Brief Title: Mesenchymal Stromal Cells for Acute Graft Versus Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: R.P.Herrmann (Other)
Collaborators: Royal Perth Hospital (Other)
Responsible Party: Sponsor-Investigator, R.P.Herrmann, Director, Cell and Tissue Therapies, Royal Perth Hospital, Royal Perth Hospital
Organization: Royal Perth Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/128; CTN 2012/0174 (Other: Therapeutics Goods Administration, Government of Australia)
Record Dates: First submitted 2012-04-26; First posted 2012-05-02 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Acute GVH Disease
Keywords: Acute graft versus host disease; Bone marrow transplantation; Mesenchymal stromal cells
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stromal cell therapy (Experimental): Mesenchymal stromal cell therapy in addition to corticosteroid therapy
  Interventions: Biological: Mesenchymal stromal cell therapy
- Corticosteroid therapy (Active Comparator)
  Interventions: Biological: Mesenchymal stromal cell therapy

INTERVENTIONS:
Biological: Mesenchymal stromal cell therapy — One arm will be randomised to receive mesenchymal stromal cell therapy in addition to corticosteroid therapy
  Other Names: Methylprednisolone; Mesenchymal stem cells

SUMMARY:
A randomised study of corticosteroid therapy with or without mesenchymal stromal cell therapy for newly diagnosed acute graft versus host disease after bone marrow transplantation or donor lymphocyte therapy.

It is hypothesised that mesenchymal stromal cell therapy will be superior

DETAILED DESCRIPTION:
Patients with newly diagnosed untreated acute graft versus host disease grades 2-4 will receive methylprednisolone 2.5mg/kg intravenously and randomised to receive or not receive allogeneic human mesenchymal stromal cells 2X10E6 intravenously on two occasions at weekly intervals

ELIGIBILITY:
Inclusion Criteria:

* Grades 2-4 acute graft versus host disease after bone marrow transplantation up to day +180 after transplantation
* Age 18-55 years

  * Must be receiving a calcineurin inhibitor

Exclusion Criteria:

* Failure to sign informed consent
* Corticosteroid therapy for 72 hours or greater
* ECOG score equal to or greater than 3

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Survival at one year after onset of graft versus host disease | One year

SECONDARY OUTCOMES:
Response at 14 days after commencement of treatment for acute graft versus host disease | 14 days
Response at 28 days after commencement of treatment of acute graft versus host disease | 28 days
Incidence of severe infection | One year
Disease free survival at one year | One year
Time to treatment failure, requiring salvage therapy | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Purtill, MB, BS, Principal Investigator — Royal Perth Hospital
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia